CLINICAL TRIAL: NCT02461511
Title: Impact Des Actions d'éducation thérapeutique Mises en Place Dans le Cadre d'un Programme autorisé auprès de Patients diabétiques hospitalisés
Brief Title: Impact of Therapeutic Education, Being Set up Under the Authorized Program for Diabetics Patients in Hospital
Acronym: ImETh
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Hôpital Léon Bérard (Other)
Responsible Party: Sponsor
Other Study IDs: Protocole#5-Version1.0
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Complications
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Therapeutic Education + Documentation: diabetic patient hospitalized patient particpating in therapeutic education program
  Interventions: Other: Therapeutic Education
- No Therapeutic Education No Documents: diabetic patient hospitalized patient without therapeutic education program no documentation submitted
- Documentation, No Therapeutic Education: diabetic patient hospitalized patient without therapeutic education program documentation submitted

INTERVENTIONS:
Other: Therapeutic Education — participation in a therapeutic education program on diabetes
  Groups: Therapeutic Education + Documentation

SUMMARY:
To Assess the impact of therapeutic education on:

* the occurrence of long term diabetes complications .
* balance of his diabetes

DETAILED DESCRIPTION:
evaluation of the benefits of therapeutic education by:

* glycated hemoglobin assay
* telephone monitoring
* quiz
* monitoring of adverse event related to diabete

ELIGIBILITY:
Inclusion Criteria: Patients

* diabetic
* hospitalized in Léon Berard
* with telephone line
* written consent given
* belong to a social security system

Exclusion Criteria:

* no diabetics
* patient having alredy completing a therapeutic education program
* minor patient (<18 years)
* pregnant woman
* without telephone line
* no belong to a social security system
* patient alredy inclued on clinical study.
* patient tutelage or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetics hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin measure | 3 months
  blood sample

SECONDARY OUTCOMES:
hopitalization | 3 months
  hospitlization related to diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Alkassoum Sapha, Medecin, Principal Investigator — medecin